CLINICAL TRIAL: NCT01106781
Title: A Non-interventional Survey on the Epidermal Growth Factor Receptor (EGFR) Mutation Status in Completely Resected Chinese Non-Small Cell Lung Cancer (NSCLC) Patients With Adenocarcinoma Histology
Brief Title: A Non-interventional Survey on the EGFR (Epidermal Growth Factor Receptor) Mutation Status in Completely Resected Chinese Non-Small Cell Lung Cancer (NSCLC) Patients With Adenocarcinoma Histology
Acronym: ICAN
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OCN-DUM-2009/1
Record Dates: First submitted 2010-04-14; First posted 2010-04-20 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: EGFR mutation test; NSCLC; Non-Interventional Study; EGFR mutation status
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Patients in this group should be histological confirmed adenocarcinoma of the lung, have received complete resection and tested for EGFR mutation.

SUMMARY:
This is a descriptive observational study. The primary objective is to explore the EGFR gene mutation status in early stage NSCLC with adenocarcinoma histology after complete resection. The patients should be histological confirmed adenocarcinoma of the lung, have received complete resection and tested for EGFR mutation in regular medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosed as adenocarcinoma type of non-small cell lung cancer
* Have completed lung cancer operation
* The tumour EGFR gene mutation status test was performed as regular medical practice

Exclusion Criteria:

* Patients who disagree to participate this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Thoracic surgery department
Sampling Method: Non-Probability Sample
Enrollment: 591 (Actual)
Dates: Start 2010-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
type and prevalence of EGFR mutation | up to 3 months

SECONDARY OUTCOMES:
Operation type and adjuvant treatment type | up to 3 months
Disease Free Survival rate | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Atkin, Study Director — Astrazeneca China R&D; Wu Yilong, Principal Investigator — Guangdong Provincial People's Hospital
Locations (13):
- China (13):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Wuhan, Hubei
  - Research Site, Nanjing, Jiangsu
  - Research Site, Suzhou, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Shenyang, Liaoning
  - Research Site, Qingdao, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Hangzhou, Zhejiang